CLINICAL TRIAL: NCT07146178
Title: Long-term Follow-up of Bio-signals and Quality of Recovery Following Implementation of Enhanced Recovery After Surgery(ERAS) Program
Brief Title: Long-term Follow-up of Bio-signals and Quality of Recovery Following Implementation of ERAS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wonju Severance Christian Hospital (Other)
Collaborators: Ministry of Trade, Industry & Energy, Republic of Korea (Other Government)
Responsible Party: Principal Investigator, Song Seung Woo, Assistant professor, Wonju Severance Christian Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ERAS2025
Record Dates: First submitted 2025-07-31; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Gynecologic Surgery; General Anesthesia
Keywords: Enhanced recovery after surgery; bio-signal monitoring
MeSH Terms: interventions — Enhanced Recovery After Surgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ERAS (Experimental)
  Interventions: Procedure: Enhanced Recovery After Surgery
- Conventional (Active Comparator)
  Interventions: Procedure: Usual Care

INTERVENTIONS:
Procedure: Enhanced Recovery After Surgery — 1. Before surgery
     * Sips of water until 6 AM on the day of surgery, followed by a 200 mL carbohydrate drink
     * Pre-emptive oral analgesics (celecoxib 200mg 1 cap + acetaminophen 650mg 2 tab)
  2. During surgery
     * Total intravenous anesthesia
     * Local anesthetic infiltration at the laparoscopic port site for post-operative pain control
  3. After surgery
     * Sips of water and a foley catheter removal on ward arrival
     * Soft meal 4 housr after surgery
     * General diet 8 hours after surgery
  Other Names: ERAS
  Arms: ERAS
Procedure: Usual Care — 1. Before surgery
     * Midnight NPO
     * No pre-emptive analgesics
  2. During surgery
     * Balanced anesthesia
  3. After surgery
     * Sips of water 8 hours after arrival in the ward
     * Foley catheter removal one day after the surgery
     * Soft meal after gas out
     * General diet after one soft meal
  Arms: Conventional

SUMMARY:
The goal of this clinical trial is to evaluate the effect of an Enhanced Recovery After Surgery(ERAS) protocol in patients undergoing gynecologic laparoscopic surgery under general anesthesia. The main question it aims to answer is: Does the ERAS protocol improve the quality of recovery compared to standard treatments?

Researchers will compare ERAS protocol with standard treatment to see if ERAS protocol improves the quality of recovery after surgery.

Participants will:

* Receive ERAS protocol during the hospitalization
* Undergo bio-signal monitoring for one month using Hi-Cardi Plus device and Galaxy Watch 7
* Visit the hospital at one week and one month after discharge
* Complete questionnaires(QOR-15K, WHO-DAS 2.0, EQ-5D-3L) at 24 hours after surgery, at discharge, one week after discharge, and one month after discharge

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 70 years
* Scheduled to undergo gynecologic laparoscopic surgery under general anesthesia
* Use of an Android smartphone

Exclusion Criteria:

* American Society of Anesthesiologists(ASA) physical status classification IV or higher
* Body Mass Index (BMI) 35 or higher
* Presence of diabetic autonomic neuropathy
* History of esophageal hiatal hernia or delayed stomach discharge
* Known allergy to local anesthesia
* Participantion in other trials that may affect study outcomes
* Inability to complete questionnaires (e.g., due to cognitive impairment)

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Quality of Recovey-15, Korean version (QoR-15K) | on 24 hours postoperatively
  This patient-reported outcome measure consists of 15 items. Each item is rated on an 11-point Likert scale (0-10), yielding a total score ranging from 0 (very poor recovery) to 150 (excellent recovery). Higher scores indicate a better postoperative recovery.
Quality of Recovey-15, Korean version (QoR-15K) | one week after hospital discharge
  This patient-reported outcome measure consists of 15 items. Each item is rated on an 11-point Likert scale (0-10), yielding a total score ranging from 0 (very poor recovery) to 150 (excellent recovery). Higher scores indicate a better postoperative recovery.
Quality of Recovey-15, Korean version (QoR-15K) | one month after hospital discharge
  This patient-reported outcome measure consists of 15 items. Each item is rated on an 11-point Likert scale (0-10), yielding a total score ranging from 0 (very poor recovery) to 150 (excellent recovery). Higher scores indicate a better postoperative recovery.
The World Health Organization Disability Assessment Schedule, 2nd Edition (WHODAS 2.0) | on 24 hours postoperatively
  WHODAS 2.0 questionnaire consists of 36 items rated on a 5-point Likert scale (1-5), yielding a total score ranging from 36 to 180. Higher scores represent greater disability and poorer functioning.
The World Health Organization Disability Assessment Schedule, 2nd Edition (WHODAS 2.0) | one week after hospital discharge
  WHODAS 2.0 questionnaire consists of 36 items rated on a 5-point Likert scale (1-5), yielding a total score ranging from 36 to 180. Higher scores represent greater disability and poorer functioning.
The World Health Organization Disability Assessment Schedule, 2nd Edition (WHODAS 2.0) | one month after hospital discharge
  WHODAS 2.0 questionnaire consists of 36 items rated on a 5-point Likert scale (1-5), yielding a total score ranging from 36 to 180. Higher scores represent greater disability and poorer functioning.
EuroQol 5-Dimension, 3-Level questionnaire (EQ-5D-3L) | on 24 hours postoperatively
  EQ-5D-3L questionnaire assesses health-related quality of life across five domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each domain is rated on a 3-level scale (1 = no problems, 2 = some problems, 3 = extreme problems), where higher scores within each domain indicate worse health status.
EuroQol 5-Dimension, 3-Level questionnaire (EQ-5D-3L) | 1 week after hospital discharge
  EQ-5D-3L questionnaire assesses health-related quality of life across five domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each domain is rated on a 3-level scale (1 = no problems, 2 = some problems, 3 = extreme problems), where higher scores within each domain indicate worse health status.
EuroQol 5-Dimension, 3-Level questionnaire (EQ-5D-3L) | 1 month after hospital discharge
  EQ-5D-3L questionnaire assesses health-related quality of life across five domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each domain is rated on a 3-level scale (1 = no problems, 2 = some problems, 3 = extreme problems), where higher scores within each domain indicate worse health status.

SECONDARY OUTCOMES:
Pain (Visual analogue scale) | on 24 hours postoperatively
  The Visual Analogue Scale (VAS) for pain ranges from 0 to 100, where 0 represents no pain and 100 represents the worst imaginable pain. Higher scores indicate more severe pain.
Pain (Visual analogue scale) | 1 week after hospital discharge
  The Visual Analogue Scale (VAS) for pain ranges from 0 to 100, where 0 represents no pain and 100 represents the worst imaginable pain. Higher scores indicate more severe pain.
Pain (Visual analogue scale) | 1 month after hospital discharge
  The Visual Analogue Scale (VAS) for pain ranges from 0 to 100, where 0 represents no pain and 100 represents the worst imaginable pain. Higher scores indicate more severe pain.
Length of stay | throughout hospitalization, expected to be 2-3 days
Total in-hospital opioid consumption | throughout hospitalization, expected to be 2-3 days
  opioid consumption to alleviate pain; exclude intraoperative remifentanil
Complication | From enrollment to one month after discharge
Readmission | From enrollment to one month after discharge
  All-cause hospital readmission within 30 days after discharge, defined as any unplanned inpatient admission to any hospital

OTHER OUTCOMES:
Heart rate variability | From discharge day to one month after discharge
  measured from wearable electrocardiography and a smart watch

CONTACTS AND LOCATIONS:
Locations (1):
- Wonju Severance Christian Hospital, Wŏnju, Gangwon-do, South Korea

IPD SHARING:
Plan to Share IPD: No